CLINICAL TRIAL: NCT06708728
Title: Study of the Etiology, Clinical Features and Short Term Outcome of Acquired Hemolytic Anemia in Hospitalized Adult Patients with Non-Neoplastic Disease
Brief Title: Study of Acquired Hemolytic Anemia in Adult Hospitalized Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Mahmoud, resident doctor, Sohag University
Other Study IDs: AEMahmoud
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood samples — blood samples for CBC parameters , peripheral blood smear, bilirubin levels and kidney function tests

SUMMARY:
the goal of the study is to identify the most common etiological factors and analyze the clinical presentations and laboratory findings in hospitalized patients with acquired hemolytic anemia associated with non-neoplastic diseases.

And to evaluate short-term outcomes, including morbidity and mortality rates, and to determine correlations between specific etiological factors and patient outcomes in these cases.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Patients diagnosed with acquired hemolytic anemia.
* Patients must be hospitalized in the Internal Medicine department at the time of diagnosis of acquired hemolytic anemia during the study period
* Patients (or their legal representatives) must provide informed

Exclusion Criteria:

* Patients with underlying neoplastic diseases.
* Patients with hereditary hemolytic anemia.
* Patients or their representatives who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in Internal Medicine department and Intermediate care unit at sohag university hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
intensive care unit admission of the patients due to progression of the disease complications. | through study completion, an average of 6 months
  Primary outcome will be ICU admission due to progression of the disease complications.

SECONDARY OUTCOMES:
mortality within duration of hospital admission | through study completion, an average of 6 months
  Secondary outcome will be mortality within duration of hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt